CLINICAL TRIAL: NCT00002825
Title: A PHASE II STUDY OF DOCETAXEL (TAXOTERE) (NSC# 628503) IN CHILDREN WITH RECURRENT SOLID TUMORS
Brief Title: Docetaxel in Treating Children With Recurrent Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02247; CCG-0962; CDR0000065008 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-03-01 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2006-05

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma; Sarcoma
Keywords: recurrent childhood rhabdomyosarcoma; recurrent neuroblastoma; recurrent osteosarcoma; recurrent childhood soft tissue sarcoma; recurrent childhood brain stem glioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Sarcoma; Osteosarcoma; Astrocytoma; Medulloblastoma; Neuroectodermal Tumors, Primitive, Peripheral; Familial ependymoma | interventions — Filgrastim; Docetaxel

ARMS (1):
- Arm I (Experimental): All patients receive docetaxel with G-CSF every 21 days for up to 12 courses.
  Interventions: Biological: filgrastim; Drug: docetaxel

INTERVENTIONS:
Biological: filgrastim
Drug: docetaxel

SUMMARY:
Phase II trial to study the effectiveness of docetaxel in treating children with recurrent solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate to docetaxel in children with recurrent sarcomas, neuroblastomas, or brain tumors.

II. Describe the toxic effects of docetaxel in these patients.

OUTLINE:

All patients receive docetaxel with G-CSF every 21 days for up to 12 courses. Patients are followed for survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically verified (at original diagnosis) solid tumor that is relapsed or refractory The following histologies are eligible:
* Sarcomas: Rhabdomyosarcoma Ewing's sarcoma, Peripheral neuroectodermal tumor (PNET), Osteosarcoma, Other soft tissue sarcomas
* Brain tumors: Ependymoma Primitive neuroectodermal tumor (PNET), High grade astrocytoma, Brain stem glioma (histologic verification not required), Neuroblastoma
* Measurable disease that can be followed clinically or radiologically required
* The following not considered measurable: Bone lesions measured by bone scan or bone marrow involvement
* Central nervous system disease documented by cerebrospinal fluid cytology
* Pleural effusion

PATIENT CHARACTERISTICS:

* Age: 21 and under at original diagnosis
* Performance status: 0-3
* Life expectancy: Greater than 2 months
* In the absence of marrow involvement:
* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 100,000/mm3 (transfusion independent)
* Hemoglobin at least 9.0 g/dL (transfusion allowed)
* With bone marrow involvement:
* Absolute neutrophil count at least 750/mm3
* Red cell and platelet support possible
* Bilirubin normal
* ALT/AST less than 1.5 times normal
* Alkaline phosphatase less than 2.5 times normal
* Creatinine no greater than 1.5 times normal OR creatinine clearance or radioisotope glomerular filtration rate at least 60 mL/min
* Not pregnant or nursing
* Adequate contraception required of fertile women

PRIOR CONCURRENT THERAPY:

* Prior bone marrow transplantation allowed:
* Must have stable engraftment without need for significant blood product support or cytokine therapy
* No concurrent immunomodulating agents
* No prior paclitaxel or docetaxel At least 2 weeks since chemotherapy (4 weeks since nitrosoureas)
* No other concurrent cancer chemotherapy
* Concurrent corticosteroids allowed for intracranial pressure in brain tumor patients provided patient has been stable for at least 4 weeks
* Corticosteroids allowed as pretreatment for docetaxel
* At least 2 months since extensive radiotherapy, defined as:
* Craniospinal Volume greater than 50% of abdominopelvic cavity
* Volume greater than one third of lung volume
* No concurrent radiotherapy
* No more than 2 prior therapies and fully recovered

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 1997-01; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Zwerdling, MD, Study Chair — University of California, Davis
Locations (36):
- United States (33):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Kaiser Permanente Medical Center-Sacramento, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Background] Blaney SM, Seibel NL, O'Brien M, Reaman GH, Berg SL, Adamson PC, Poplack DG, Krailo MD, Mosher R, Balis FM. Phase I trial of docetaxel administered as a 1-hour infusion in children with refractory solid tumors: a collaborative pediatric branch, National Cancer Institute and Children's Cancer Group trial. J Clin Oncol. 1997 Apr;15(4):1538-43. doi: 10.1200/JCO.1997.15.4.1538. PMID 9193350
- [Result] Zwerdling T, Krailo M, Monteleone P, Byrd R, Sato J, Dunaway R, Seibel N, Chen Z, Strain J, Reaman G; Children's Oncology Group. Phase II investigation of docetaxel in pediatric patients with recurrent solid tumors: a report from the Children's Oncology Group. Cancer. 2006 Apr 15;106(8):1821-8. doi: 10.1002/cncr.21779. PMID 16532433